CLINICAL TRIAL: NCT04801784
Title: Hemodynamic-guided Fluid Balance Neutralization During Continuous Renal Replacement Therapy in Critically Ill Patients: the GO NEUTRAL Randomized Controlled Multi-center Study
Brief Title: Fluid Balance Neutralization During CRRT (Continuous Renal Replacement Therapy)
Acronym: GO-NEUTRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69HCL20_1243; 2021-A00692-39 (Other: ANSM)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fluid Overload
Keywords: Fluid Overload; fluid balance; continuous renal replacement therapy; net ultrafiltration; acute kidney injury; hemodynamic monitoring; preload dependence; hemodynamic instability; acute circulatory failure; shock; deresuscitation
MeSH Terms: conditions — Edema; Acute Kidney Injury; Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Group allocation masking to staff performing result analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid balance neutralization (Experimental): Fluid balance neutralization using increased net ultrafiltration, aiming to neutralize the cumulative fluid input received over the first 72 hours of study participation.
  Interventions: Procedure: Increased net ultrafiltration with advanced hemodynamic monitoring
- Standard care (Active Comparator): Active control group of positive fluid balance during the first 72 hours of study participation with zero or near-zero net ultrafiltration.
  Interventions: Procedure: Zero or near-zero net ultrafiltration

INTERVENTIONS:
Procedure: Increased net ultrafiltration with advanced hemodynamic monitoring — A net ultrafiltration rate of 100 ml/h or more will be applied during the first 72 hours of study participation. To insure the hemodynamic security of the intervention, it is associated with an advanced hemodynamic monitoring protocol which encompasses cardiac index, preload dependence assessment (using postural maneuvers), lactate levels and central venous pressure evaluation. The hemodynamic monitoring protocol allows the decrease or suspension of the neutral ultrafiltration rate in case of hemodynamic instability or of hemodynamic status considered at risk of worsening if net ultrafiltration rate is maintained.
  Arms: Fluid balance neutralization
Procedure: Zero or near-zero net ultrafiltration — The active control group aims to represent the present standard of care of net ultrafiltration management in the first 72 hours of study participation in patients with critical illness. This will be performed by setting the net ultrafiltration rate to 0 up to 25 ml/h.
  Arms: Standard care

SUMMARY:
Fluid overload is associated with increased mortality in critically ill patients with acute kidney injury. Fluid balance controlled is associated with improved outcome in observational studies, and is deemed safe in interventional trials.

The objective of the study is to keep fluid balance neutral by matching the net ultrafiltration rate to fluid inputs in patients with vasoplegia, and treated with continuous renal replacement therapy (CRRT), while insuring its security using advanced hemodynamic monitoring with continuous cardiac output monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 yo or more, affiliated to a social security system
* Treated with vasopressors for acute circulatory failure
* With KDIGO stage 3 acute kidney injury
* Treated with continuous renal replacement therapy for less than 24 jours
* Monitored with a calibrated continuous cardiac output device

Exclusion Criteria:

* Treatment by ECMO (extracorporeal membrane oxygenation)
* Active hemorrhage necessitating transfusion
* Maintenance dialysis or renal graft recipient
* Switch to intermittent hemodialysis is scheduled in the next 72 hours
* Acute cerebral stroke complicated by coma and under mechanical ventilation
* Acute fulminant hepatitis
* Postural maneuver (passive leg raising or Trendelenburg) cannot be performed (amputation, inferior vena cava obstruction)
* Pregnancy or lactating
* Withdrawal or limitation of care
* Moribund patient
* Patient under protective measures/wardship
* Inclusion in another trial whose main outcome is cumulative fluid balance, or whose intervention targets hemodynamic physiology, fluid balance or net ultrafiltration.
* Patient previously enrolled in the same study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Cumulative fluid balance | 72 hours from study inclusion (H72)
  The cumulative fluid balance (in ml) will be calculated as the total amount of input received by the patients (including IV fluids and medications, blood products, hydration and nutrition), minus the total output over the same period of time (including urine output, net ultrafiltration, and drains). The cumulative fluid balance at H72 will be compared between study groups in alive patients at H72.

SECONDARY OUTCOMES:
Number of hemodynamic episodes | 72 hours from study inclusion
  Hemodynamic instability is defined as the appearance of mottles, a mean arterial pressure < 65 mm Hg and requiring urgent intervention, a decrease in cardiac index > 15%, or tachycardia > 120 beats per minute (bpm).
Number of hemodynamic episodes with preload dependence status | 72 hours from study inclusion
  Hemodynamic episodes defined as stated above, that were associated with preload dependence, defined as a significant increase in cardiac index when performing a postural maneuver. This test will be performed every 4 hours as part of the hemodynamic protocol
Number of Major Adverse Kidney Events (MAKE) | 90 days from study inclusion
  MAKE is a composite criterion applied to participants, composed of either the persistence of renal impairment at Day90 (defined as a serum creatinine > 2 x baseline value), renal replacement therapy dependence at Day90, or death at Day90. A separate analysis of each components of the MAKE 90 outcome will be performed.
Mean arterial pressure | Every 4 hours from inclusion to 72 hours after inclusion
  Repeated measurement or assessment of mean arterial pressure, cardiac index, lactatemia, and vasopressor dose will make it possible to assess the hemodynamic effect of study intervention
Cardiac index | Every 4 hours from inclusion to 72 hours after inclusion
  Repeated measurement or assessment of mean arterial pressure, cardiac index, lactatemia, and vasopressor dose will make it possible to assess the hemodynamic effect of study intervention
Lactatemia | Every 4 hours from inclusion to 72 hours after inclusion
  Repeated measurement or assessment of mean arterial pressure, cardiac index, lactatemia, and vasopressor dose will make it possible to assess the hemodynamic effect of study intervention
Vasopressor dose administered | Every 4 hours from inclusion to 72 hours after inclusion
  Repeated measurement or assessment of mean arterial pressure, cardiac index, lactatemia, and vasopressor dose will make it possible to assess the hemodynamic effect of study intervention
Cumulative fluid balance | 24 hours and day 7 from study inclusion
  The cumulative fluid balance will be calculated as stated for the primary outcome at Hours24. It will be estimated using body weight variation between inclusion and day 7.
Cumulative net ultrafiltration | 24 hours, 72 hours and day 7 from study inclusion
  The cumulative net ultrafiltration is reported by CRRT (continuous renal replacement therapy) generators ad collected every 4 hours from inclusion to 72 hours after inclusion.
Number of respiratory and circulatory failure free days | Day 28 of study inclusion
  Organ failure free days are defined as the number of days without organ support, and censored at 28 days of inclusion. Weaning of mechanical ventilation is defined as being free of IMV for 48 hours or more. Weaning of vasopressor is defined as being free of any vasopressor administration for 48 hours or more. Participant who die are over the 28-day period are assigned a value of 0 organ failure free days.
Severity of organ failures using the SOFA score | from inclusion to 72 hours of study inclusion
  Organ failure severity is quantified using the SOFA score (Sepsis-related organ failure assessment), and is collected at inclusion, and daily until Hours 72. The SOFA score assesses 6 physiological systems: respiratory, circulatory, coagulation, liver, renal and neurological.
PaO2/FiO2 ratio | 24 hours, 48 hours, and 72 hours from study inclusion
  Intensity of pulmonary hydrostatic edema will be quantified using the PaO2/FiO2 ratio variation from inclusion to Hours24, Hours48 and Hours72 of study inclusion
Extravascular lung water index | 24 hours, 48 hours, and 72 hours from study inclusion
  Intensity of pulmonary hydrostatic edema will be quantified using the extravascular lung water index reported by the continuous cardiac monitoring device, from inclusion to Hours24, Hours48 and Hours72 of study inclusion
Hospitalisation duration | Day 90 of study inclusion
  Hospitalisation duration will be quantified as the delay between participant admission and discharge from hospital, censored at day 90 from inclusion.
Duration of stay in Intensive Care Unit (ICU) | Day 90 of study inclusion
  Duration of stay in ICU will be quantified as the delay between participant admission and discharge from ICU, censored at day 90 from inclusion
Survival | Day 28 and 90 of study inclusion
  Vital status (death/alive) will be reported at D28 and D90 of study inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BITKER, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Bitker L, Pradat P, Dupuis C, Klouche K, Illinger J, Souweine B, Richard JC. Fluid balance neutralization secured by hemodynamic monitoring versus protocolized standard of care in critically ill patients requiring continuous renal replacement therapy: study protocol of the GO NEUTRAL randomized controlled trial. Trials. 2022 Sep 22;23(1):798. doi: 10.1186/s13063-022-06735-6. PMID 36138465